CLINICAL TRIAL: NCT03001427
Title: Neurocognition, Lifestyle Modification, and Treatment Resistant Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00055703_1
Record Dates: First submitted 2016-12-20; First posted 2016-12-23 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Treatment-Resistant Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structured center-based lifestyle intervention (Experimental): The Structured center-based Lifestyle Intervention (C-LIFE) will include individualized plans for the DASH diet, weight management, and aerobic exercise.
  Interventions: Behavioral: Structured center-based lifestyle intervention
- Standard education and physician advice (Experimental): The Medical Management with Standardized Education and Physician Advice (SEPA) will consist of encouragement to achieve an ideal body weight and engage in exercise as part of routine counseling in primary care, but no special program will be delivered to enhance the participants' ability to comply with these recommendations.
  Interventions: Behavioral: Standard education and physician advice

INTERVENTIONS:
Behavioral: Structured center-based lifestyle intervention
  Arms: Structured center-based lifestyle intervention
Behavioral: Standard education and physician advice
  Arms: Standard education and physician advice

SUMMARY:
This application proposes to extend an ongoing NHLBI clinical trial (NCT02342808) examining the efficacy of a lifestyle intervention combining the Dietary Approaches to Stop Hypertension (DASH) diet with caloric restriction and aerobic exercise to lower and control BP in individuals with RH. In the parent trial, participants with RH will be randomized to either: (1) a 4-month adjunctive lifestyle intervention designed to lower BP through exercise and diet (C-LIFE), or; (2) a standardized education and physician advice (SEPA) control condition.

The current protocol will collect additional assessments of neurocognition (executive function, processing speed, and memory), endothelial function (brachial artery flow-mediated dilation), and cerebrovascular reserve (a measure of prefrontal cortex tissue oxygenation) in 120 participants at baseline, following completion of the 4-month intervention, and again after one year, in order to examine neurocognitive improvements and their potential mediators.

ELIGIBILITY:
Inclusion Criteria:

* Documented resistant hypertension (RH). In the absence of a specific RH diagnosis, individuals being treated for two or more weeks with 3 antihypertensive medications of different classes, including a diuretic if tolerated, with clinic SBP ≥ 130 mm Hg or DBP ≥ 80 mm Hg, will be eligible. Individuals being treated with 4 or more antihypertensive medications, including a diuretic if tolerated, with SBP ≥ 120 or DBP ≥ 80 mm Hg will also be eligible.
* Adherent to prescribed medications
* Overweight (BMI ≥ 25 kg/m2)
* Sedentary
* Willing to be randomized to one of the 2 treatment groups and able to fully participate in intervention
* Informed consent

Exclusion Criteria:

* Secondary HTN, non-adherence to anti-HTN medications
* Severe CKD (eGFR <40 ml/min/1.73m2)
* Severe ischemic heart disease (CCS Class 3 or 4 angina or evidence of ischemia at <85% heart rate reserve on treadmill testing)
* Severe heart failure (NYHA association Class 3 or 4), high grade arrhythmias, severe valvular heart disease
* Severe asthma or chronic obstructive lung disease
* Diabetes requiring insulin
* Musculoskeletal or neurologic problems that would preclude participation in aerobic exercise training
* Major psychiatric disorder, a history of drug abuse, alcohol consumption >14 drinks/week
* Life-limiting comorbid medical condition such as cancer
* Prior gastric bypass surgery
* Currently pregnant
* Cognitively impaired

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Executive Function composite | Baseline to immediate post-treatment (4 months)
  Trail Making Test Part B, Stroop Color-Word Section, Animal Naming, COWA, CVLT-II Discrimination Index
Processing Speed composite | Baseline to immediate post-treatment (4 months)
  Trail Making Test Part A, Stroop Word Section, Stroop Color Section, Digit Symbol, Ruff 2&7 Test
Memory composite | Baseline to immediate post-treatment (4 months)
  CVLT-II Learning, CVLT-II Free Recall, RCFT Recall, Digit Spa

SECONDARY OUTCOMES:
Brachial Artery Flow-Mediated Dilation | Baseline to immediate post-treatment (4 months)
Prefrontal Cortex Tissue Oxygenation Index | Baseline to immediate post-treatment (4 months)

OTHER OUTCOMES:
Executive Function composite | Baseline to follow-up (1 year)
  Trail Making Test Part B, Stroop Color-Word Section, Animal Naming, COWA, CVLT-II Discrimination Index
Processing Speed composite | Baseline to follow-up (1 year)
  Trail Making Test Part A, Stroop Word Section, Stroop Color Section, Digit Symbol, Ruff 2&7 Test
Memory composite | Baseline to follow-up (1 year)
  CVLT-II Learning, CVLT-II Free Recall, RCFT Recall, Digit Spa

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumenthal JA, Sherwood A, Smith PJ, Mabe S, Watkins L, Lin PH, Craighead LW, Babyak M, Tyson C, Young K, Ashworth M, Kraus W, Liao L, Hinderliter A. Lifestyle modification for resistant hypertension: The TRIUMPH randomized clinical trial. Am Heart J. 2015 Nov;170(5):986-994.e5. doi: 10.1016/j.ahj.2015.08.006. Epub 2015 Aug 14. PMID 26542509